CLINICAL TRIAL: NCT01933360
Title: Sublingual Versus Vaginal Misoprostol for Cervical Dilatation 1 or 3 Hours Prior to Surgical Abortion
Brief Title: Misoprostol for Cervical Priming Prior to Vacuum Aspiration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W500M
Record Dates: First submitted 2013-08-25; First posted 2013-09-02 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: First Trimester Pregnancy; Surgical Termination of Pregnancy
Keywords: Misoprostol; First trimester pregnancy; Surgical abortion; Cervical priming
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Misoprostol sublingual,1h (Active Comparator): Administration of misoprostol sublingually 1h prior to surgery
  Interventions: Drug: Misoprostol sublingual, 1h; Drug: Placebo vaginal, 1h
- Misoprostol sublingual. 3h (Active Comparator): Administration of misoprostol sublingually 3h prior to surgery
  Interventions: Drug: Misoprostol sublingual, 3h; Drug: Placebo vaginal, 3h
- Misoprostol vaginal,1h (Active Comparator): Administration of misoprostol vaginally 1h prior to surgery
  Interventions: Drug: Placebo sublingual,1h; Drug: Misoprostol vaginal, 1h
- Misoprostol vaginal,3h (Active Comparator): Administration of misoprostol vaginally 3h prior to surgery
  Interventions: Drug: Misoprostol vaginal, 3h; Drug: Placebo sublingual, 3h

INTERVENTIONS:
Drug: Misoprostol sublingual, 1h — Misoprostol is administered sublingually 1 hour prior to surgical termination of early pregnancy
  Other Names: Misoprostol (Cytotec)
  Arms: Misoprostol sublingual,1h
Drug: Placebo sublingual,1h — Placebo for misoprostol is administered sublingually 1 hour prior to surgical termination of early pregnancy
  Arms: Misoprostol vaginal,1h
Drug: Misoprostol sublingual, 3h — Misoprostol is administered sublingually, 3 hours prior to surgical termination of early pregnancy
  Arms: Misoprostol sublingual. 3h
Drug: Misoprostol vaginal, 1h — Misoprostol is administered vaginally 1 hour prior to surgical termination of early pregnancy
  Arms: Misoprostol vaginal,1h
Drug: Misoprostol vaginal, 3h — Misoprostol is administered vaginally 3 hours prior to surgical termination of early pregnancy
  Arms: Misoprostol vaginal,3h
Drug: Placebo sublingual, 3h — Placebo for misoprostol is administered sublingually 3 hours prior to surgical termination of early pregnancy
  Arms: Misoprostol vaginal,3h
Drug: Placebo vaginal, 1h — Placebo for misoprostol is administered vaginally 1 hour prior to surgical termination of early pregnancy
  Arms: Misoprostol sublingual,1h
Drug: Placebo vaginal, 3h — Placebo for misoprostol is administered vaginally 3 hours prior to surgical termination of early pregnancy
  Arms: Misoprostol sublingual. 3h

SUMMARY:
Despite of the widespread use, and extensive studies, the optimal route of administration of misoprostol before surgical abortion remains to be defined. Following administration of 400 mcg vaginally as per clinical guidelines, the time for optimal priming seems to be 3 hours, but the longer the interval the greater the risk or bleeding and expulsion of the uterine contents before the surgical evacuation. Sublingual administration seems to give adequate plasma concentration and cervical priming faster than oral or vaginal administration. This may allow a shorter waiting time with maintained efficacy, less side effects and logistic advantages.

ELIGIBILITY:
Inclusion Criteria:

* women opting for first trimester surgical abortion
* nulliparous
* able and willing to provide informed consent

Exclusion Criteria:

* unwilling to participate,
* unable to communicate in Swedish and English and
* minors (i.e. women < 18 years of age),
* contraindications to misoprostol
* women with pathological pregnancies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Force needed for cervical dilatation | Measured at surgery
  Cervical dilation is evaluated at surgery using Hulka dilators connected to a tonometer. Force and time needed for the dilatation is recorded by the tonometer

SECONDARY OUTCOMES:
Cervical diameter | Measured at surgery
  Cervical dilation is evaluated at surgery using Hulka dilators connected to a tonometer.The largest dilator that can pass through the inner cervical os without any resistance corresponds to the presurgical cervical diameter
Number of Participants with Adverse Events | Up to surgery
  Any side effects or symptoms such as nausea, vomiting, uterine cramps, expulsion, bleeding, rash, chills, blood pressure etc are recorded continuously from misoprostol administration until to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Saav I, Kopp Kallner H, Fiala C, Gemzell-Danielsson K. Sublingual versus vaginal misoprostol for cervical dilatation 1 or 3 h prior to surgical abortion: a double-blinded RCT. Hum Reprod. 2015 Jun;30(6):1314-22. doi: 10.1093/humrep/dev071. Epub 2015 Apr 2. PMID 25840429